CLINICAL TRIAL: NCT05058040
Title: A Clinical Study to Evaluate the Long-Term Safety Sodium Oligomannate Capsules
Brief Title: A Clinical Study to Evaluate the Long-Term Safety Sodium Oligomannate Capsules (GV-971)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Green Valley (Shanghai) Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GV-971-PMS-A
Record Dates: First submitted 2021-05-16; First posted 2021-09-27 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GV-971 (Experimental): The recommended dose regimen for subjects: GV-971 450 mg (3 capsules) per dose, bid, po. in morning and evening
  Interventions: Drug: Sodium Oligomannate Capsules

INTERVENTIONS:
Drug: Sodium Oligomannate Capsules — Sodium Oligomannate Capsules, each capsule contains 150 mg of sodium oligomannate. The recommended treatment is oral administration, 450 mg (3 capsules) per dose, bid, in morning and evening.

SUMMARY:
A clinical study to evaluate the long-term safety of Sodium Oligomannate Capsules (GV-971)

DETAILED DESCRIPTION:
Sodium oligomannate (Code: GV-971), a marine-derived oligosaccharide after extraction, separation and degradation from algae, can play a role in the treatment of Alzheimer's disease by reconditioning the dysbiosis of gut microbiota, preventing peripheral immune cells from invading the brain, inhibiting the inflammatory response in the brain, and targeting protein folding errors in the brain tissue. Phase I clinical study shows GV-971 was safe and tolerated in healthy adult volunteers when administered continuously at 1200 mg/dose or 1500 mg/day (750 mg/dose, bid) for 5 days. Phase II and III clinical studies show that the treatment of GV-971 at 900 mg/day dosage for 36 weeks can significantly improve the cognitive function of patients with mild to moderate Alzheimer's disease (AD) and was safe and well-tolerated.

Sodium Oligomannate Capsules obtained approval from China's National Medical Products Administration (NMPA) on November 2, 2019, with approval letter number of 2019S00571. This product is a chemical drug with a registration classification of 1.2. It is approved for the clinical indication of mild to moderate Alzheimer's disease and the function of improving the cognitive function of patients. The clinical dosage and administration is 3 capsules (450 mg)/time, bid, po.

Due to the limited number of subjects and observation period of medication in completed GV-971 clinical studies, and the screening of patients with the strict inclusion and exclusion criteria, the adverse reactions and long-term safety of GV-971 cannot be comprehensively observed and recorded. Therefore, according to the requirements of the NMPA for the marketing of new drugs, this study is intended to further carry out a post-marketing investigation on expanded population using a design of a 96-week intensive monitoring clinical trial to determine the incidence of known adverse reactions of GV-971 under long-term administration, observe the occurrence of new adverse reactions, analyze the correlation, incidence, severity, and risk factors of adverse reactions/events, and better guide the rational use of drugs in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for this study must meet all of the following criteria:

  1. ≥18 years of age;
  2. Signed informed consent form;
  3. Patients receiving GV-971 treatment prescribed by clinicians;

Exclusion Criteria:

* A subject may be excluded from participation in the study if any of the following apply:

  1. Patients who may be allergic to Sodium Oligomannate Capsules as judged by the investigator;
  2. Female participants who are pregnant or lactating;
  3. Patients who cannot cooperate to complete the follow-up inquiries;
  4. Any other diseases or conditions that are inappropriate to participate in this clinical trial in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Long-term safety of GV-971 in clinical practice during 48 weeks | Week 48
  The incidence of adverse reactions and AE/SAE in patients treated with GV-971 during the 48-week monitoring period
Long-term safety of GV-971 in clinical practice during 96 weeks | Week 96
  The incidence of adverse reactions and AE/SAE in patients treated with GV-971 during the 96-week monitoring period

SECONDARY OUTCOMES:
Safety Endpoints: Vital signs, laboratory tests , electrocardiogram, and early withdrawal from the study during 48 weeks | 48-week
  The incidence of adverse events and adverse reactions in patients with liver insufficiency and renal insufficiency receiving GV-971 during 48 weeks
Safety Endpoints: Vital signs, laboratory tests , electrocardiogram, and early withdrawal from the study during 96 weeks | 96-week
  The incidence of adverse events and adverse reactions in patients with liver insufficiency and renal insufficiency receiving GV-971 during 96 weeks

CONTACTS AND LOCATIONS:
Locations (63):
- China (63):
  - Anhui Mental Health Center, Hefei, Anhui
  - The First Affiliated Hospital of USTC(Anhui Provincial Hospital), Hefei, Anhui
  - Beijing Bo'ai Hospital, Beijing, Beijing Municipality
  - Beijing Geriatric Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Dongfang Hospital Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Sanbo Brain Hospital Capital Medical University, Beijing, Beijing Municipality
  - Chongqing 11th People's Hospital (Chongqing Special Care Hospital), Chongqing, Chongqing Municipality
  - Xiamen Xianyue Hospital, Xianmencun, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Red Cross Hospital of Guangzhou, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Luohu District People's Hospital, Shenzhen, Guangdong
  - Shenzhen Second People's Hospital (The First Affiliated Hospital of Shenzhen University), Shenzhen, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - Guihang Guiyang Hospital, Guiyang, Guizhou
  - Second People's Hospital of Guizhou Province, Guiyang, Guizhou
  - The First Affiliated Hospital of Guizhou University of Chinese Medicine, Guiyang, Guizhou
  - The Second Affiliated Hospital of Guizhou University of Chinese Medicine, Guiyang, Guizhou
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - General Hospital of North China Petroleum Administration (North China Hospital Affiliated to University of Chinese Academy of Sciences), Renqiu, Hebei
  - Wuhan Central Hospital, Wuhan, Hubei
  - Wuhan Mental Health Center, Wuhan, Hubei
  - Lianyungang Chinese Medicine Hospital, Lianyungang, Jiangsu
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nantong No.1 People's Hospital, Nantong, Jiangsu
  - Changshu No.2 People's Hospital, Suzhou, Jiangsu
  - Suzhou Guangji Hospital, Suzhou, Jiangsu
  - Suzhou Municipal Hospital(Geriatrics), Suzhou, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Suzhou Ninth People's Hospital, Suzhou, Jiangsu
  - Taizhou Second People's Hospital, Taizhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Zhenjiang mental health center, Zhenjiang, Jiangsu
  - Jinan Central Hospital Affiliated To Shandong University, Jinan, Shandong
  - Shandong Mental Health Center, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Fengxian District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai Fifth People's Hospital,Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area People's Hospital, Shanghai, Shanghai Municipality
  - Tong Ren Hospital,Shanghai Jiao Tong University School Of Medicine, Shanghai, Shanghai Municipality
  - Second hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Xi’an, Shanxi
  - Xi 'an Baoshihua Changqing Hospital, Xi’an, Shanxi
  - Xi'an Central Hospital, Xi’an, Shanxi
  - Chengdu Eighth People's Hospital, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Sichuan Baoshihua Hospital, Chengdu, Sichuan
  - Chengdu Fourth People's Hospital, Chengdu, Sichuang
  - The Fifth People's Hospital of Chengdu, Chengdu, Sichuang
  - Nanchong Central Hospital, Nanchong, Sichuang
  - Huzhou Third Municipal Hospital, Huzhou, Zhejiang
  - Huamei Hospital,University of Chinese Academy of Sciences, Ningbo, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Ningbo Kangning Hospital, Ningbo, Zhejiang
  - Wenzhou People's Hospital, Wenzhou, Zhejiang